CLINICAL TRIAL: NCT01824953
Title: Significance of Helicobacter Pylori Infection and Pepsinogen Levels on the Prognosis of Atrophic Gastritis - Observational Study
Brief Title: Long-term Follow-up Prognosis of Atrophic Gastritis After 3 Years
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sun-Young Lee, Associate professor, Konkuk University Medical Center
Other Study IDs: KUH1010393; 1010393 (Other: Konkuk University Medical Center); KUH 1010393 (Other: Konkuk University Medical Center)
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Gastric Neoplasm; Gastric Cancer; Gastric Adenoma; Gastric Atrophy; Intestinal Metaplasia
Keywords: Gastric atrophy; Helicobacter pylori; Pepsinogen; Gastric cancer; Gastric adenoma
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum for Helicobacter pylori antibody and pepsinogen levels Gastric biopsy for the diagnosis of intestinal metaplasia, atrophy, inflammatory cells, Helicobacter pylori, and the presence of gastric neoplasm if any.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- atrophy-/Hp- group: Subjects without Helicobacter pylori infection and without atrophy
- atrophy-/Hp+: Subjects with Helicobacter pylori infection and without atrophy
- atrophy+/Hp+: Subjects with Helicobacter pylori infection and with atrophy
- atrophy+/Hp-: Subjects without Helicobacter pylori infection and with atrophy

SUMMARY:
Serum pepsinogen (PG) levels are considered reliable markers for progression of atrophic gastritis with a stepwise reduction in the serum PG I level or PG I/II ratio. A combination of serum PG levels and Helicobacter pylori serology are used as a biomarker strategy for detection of individuals at increased risk of gastric neoplasm based on Correa's hypothesis. The investigators aimed to uncover whether this combination method could predict the risk of gastric neoplasms and the progression of chronic atrophic gastritis after 3 years. All the participants will be followed for an expected average of 3 years.

DETAILED DESCRIPTION:
According to the Correa's hypothesis, the combination method using serum pepsinogen levels and serum Helicobacter pylori antibody would predict the risk and cell type of gastric neoplasm. However, in endemic regions of H. pylori infection such as in East Asian countries (Korea, Japan, and China), most of the aged population are have current or had past H. pylori infection. Therefore, in this study, we are going to uncover whether the risk of gastric neoplasm is significantly higher in the atrophy(+)/H. pylori(-) group followed by atrophy(+)/H. pylori(+), atrophy(-)/H. pylori(+), and atrophy(-)/H. pylori(-) groups. In addition, we are going to investigate whether those slow-growing gastric neoplasms such as differentiated gastric cancers with Lauren's intestinal type and gastric adenoma are more commonly developed in atrophy group following the Correa's hypothesis, whereas rapid-growing gastric neoplasms such as poorly-cohesive carcinoma or undifferentiated gastric cancers with Lauren's diffuse type are more commonly developed in the subjects without atrophy. Taken as a whole, our study result will provide an evidence whether this biomarker strategy are useful for the detection of individuals at increased risk of gastric neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* Korean adults older than 18 year-old
* Subjects who agreed on serum pepsinogen tests, H. pylori serology, and upper gastrointestinal endoscopy on the same day

Exclusion Criteria:

* Subjects who had past history of gastric surgery
* Abnormal endoscopic or laboratory finding that require further treatment
* Any evidence of malignancy other than gastric neoplasm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic Korean adults who underwent serum PG tests, H. pylori serology, and upper gastrointestinal endoscopy on the same day at our center.
Sampling Method: Non-Probability Sample
Enrollment: 3328 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Newly developed gastric neoplasm | December 31, 2013
  Newly developed gastric neoplasm

SECONDARY OUTCOMES:
Degree of gastric atrophy | December 31, 2013
  Degree of gastric atrophy measured by serum pepsinogen I and II levels

OTHER OUTCOMES:
Helicobacter pylori | December 31, 2013
  Presence of Helicobacter pylori infection

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Young Lee, MD, Principal Investigator — Department of Internal Medicine, Konkuk Universtiy Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea